CLINICAL TRIAL: NCT05753618
Title: A Randomized Pragmatic Trial Evaluating Omission of Granulocyte Colony-stimulating Factors in Breast Cancer Patients Receiving Paclitaxel Portion of Dose-dense Adriamycin-cyclophosphamide and Paclitaxel Chemotherapy (REaCT-OGF)
Brief Title: Evaluating Omission of Granulocyte Colony-stimulating Factors in Breast Cancer Patients Receiving Paclitaxel Portion of Dose-dense Adriamycin-cyclophosphamide and Paclitaxel Chemotherapy
Acronym: REaCT-OGF
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REaCT-OGF
Record Dates: First submitted 2023-01-24; First posted 2023-03-03 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Early-stage Breast Cancer
Keywords: Filgrastim; Pegfilgrastim; Bone pain; Paclitaxel
MeSH Terms: conditions — Breast Neoplasms | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Receive G-CSF (Active Comparator): Receive G-CSF injections (either filgrastim or pegfilgrastim) after each cycle of paclitaxel chemotherapy.
  Interventions: Drug: Granulocyte Colony-Stimulating Factor (G-CSF)
- Omission of G-CSF (Experimental): Omission of G-CSF injections after each cycle of paclitaxel chemotherapy.
  Interventions: Drug: Omission of Granulocyte Colony-Stimulating Factor (G-CSF)

INTERVENTIONS:
Drug: Granulocyte Colony-Stimulating Factor (G-CSF) — Participants will receive G-CSF injection (either filgrastim or pegfilgrastim) after each paclitaxel cycle of DD-AC/T chemotherapy.
  Other Names: Filgrastim; Pegfilgrastim
  Arms: Receive G-CSF
Drug: Omission of Granulocyte Colony-Stimulating Factor (G-CSF) — Participants will omit the use of G-CSF (either filgrastim or pegfilgrastim) after each paclitaxel cycle of DD-AC/T chemotherapy
  Arms: Omission of G-CSF

SUMMARY:
The goal of this randomized, pragmatic clinical trial is to evaluate the omission of granulocyte colony-stimulating factors (G-CSF) in breast cancer patients receiving paclitaxel portion of dose-dense adriamycin-cyclophosphamide and paclitaxel (DD-AC/T) chemotherapy. Participants will be randomized to either take G-CSF while on the paclitaxel portion of DD-AC/T chemotherapy or to omit G-CSF while on the paclitaxel portion of DD-AC/T chemotherapy.

DETAILED DESCRIPTION:
Optimal curative chemotherapy treatment in the early-stage setting for breast cancer patients can reduce the risk of recurrence and result in improvement in breast cancer survival. The pivotal Cancer and Leukemia Group B (CALGB) 9741 clinical trial demonstrated improved efficacy from administering 4 cycles of adriamycin and cyclophosphamide (AC) followed by 4 cycles of paclitaxel using a dose-dense schedule every 2-weeks instead of every 3 weeks in patients with high-risk early-stage breast cancer. It has since become a widely accepted standard care treatment option. Granulocyte colony-stimulating factor (G-CSF) such as filgrastim (FIL) and pegfilgrastim (PEG) are key supportive medications used with the dose-dense regimen to facilitate timely recovery of neutrophil count before the next cycle of treatment. However, G-CSF is associated with increased bone pain after chemotherapy (up to 40%) and drug-induced fever, which can result in additional clinical or emergency room visits. Clinicians have questioned if primary prophylactic G-CSF use is necessary with paclitaxel in the dose-dense regimen and the risk of hematological toxicity, such as the risk of low neutrophils and the risk of infection is lower with paclitaxel. Results from two retrospective studies suggest that it is safe and feasible to omit G-CSF during the paclitaxel portion of the DD-AC/T regimen. Based on the current trial data, there is a stong suggestion that it is safe, feasible and likely preferable to omit G-CSF during the paclitaxel portion of DD-AC/T chemotherapy. Given the majority of chemotherapy dose delays are related to issues such as bone pain (from G-CSF and paclitaxel) and peripheral neuropathy (from paclitaxel), and this may even be exacerbated by the use of G-CSF, it is anticipated that omitting G-CSF during paclitaxel chemotherapy may improve completion rates while improving health related quality of life (HR-QoL). Therefore, the researchers propose a randomized study to further evaluate patient-reported bone pain and HR-QoL from the omission of primary prophylactic G-CSF use during the paclitaxel portion of DD-AC/T chemotherapy while demonstrating supportive evidence that omitting G-CSF is safe and feasible.

ELIGIBILITY:
Inclusion Criteria:

* Patients with early-stage or locally-advanced breast cancer receiving neoadjuvant or adjuvant DD-AC/T chemotherapy requiring primary febrile neutropenia prophylaxis with G-CSF
* Able to provide verbal consent
* Able to complete questionnaires in English or French

Exclusion Criteria:

* No access to pegfilgrastim or filgrastim prior to randomization
* Metastatic cancer
* Known hypersensitivity to filgrastim or pegfilgrastim or one of its components
* Patients received prior cytotoxic chemotherapy within the last 5 years
* Patients with uncontrolled inter-current illness that would limit compliance with study requirements or other significant diseases or disorders that, in the investigator's opinion, would exclude the subject from participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Patient-reported bone pain during cycle 1 of paclitaxel | At the end of cycle 1 of paclitaxel chemotherapy (each cycle is 14 days)
  The primary outcome is patient-reported bone pain from day 1 to 5 during cycle 1 of paclitaxel chemotherapy. The total measure of bone pain over the five days will be summarized by the area under the curve (AUC) using the trapezoidal quadrature method for patients reported daily pain score from day 1 to 5 during cycle 1 of paclitaxel chemotherapy. Day 1 being the morning after first dose of G-CSF injection, or 48 hours after chemotherapy injection in the No G-CSF arm. The daily pain score ranges from 0-40. Peak pain is defined as the maximum pain rating over day 1 to day 5. To reiterate the scoring system, every morning, patients are asked to rate the most severe pain they experienced in the last 24 hours on a visual analogue scale (VAS) from 0 (no pain) to 10 (pain as bad as you can imagine). The X axis of the AUC represents time (i.e., days) and the Y axis represents pain severity (0-10).

SECONDARY OUTCOMES:
Patient-reported bone pain across all paclitaxel cycles | After each of the paclitaxel chemotherapy cycles (each cycle is 14 days)
  Bone pain mean AUC across all cycles of paclitaxel chemotherapy. The total measure of bone pain over the five days will be summarized by the area under the curve (AUC) using the trapezoidal quadrature method for patients reported daily pain score from day 1 to 5 during all cycles of paclitaxel chemotherapy. Day 1 being the morning after first dose of G-CSF injection, or 48 hours after chemotherapy injection in the No G-CSF arm. The daily pain score ranges from 0-40. Peak pain is defined as the maximum pain rating over day 1 to day 5. To reiterate the scoring system, every morning, patients are asked to rate the most severe pain they experienced in the last 24 hours on a visual analogue scale (VAS) from 0 (no pain) to 10 (pain as bad as you can imagine). The X axis of the AUC represents time (i.e., days) and the Y axis represents pain severity (0-10).
Peak bone pain experienced | Days 1 to 5 of the each of the paclitaxel chemotherapy cycles (each cycle is 14 days)
  Peak bone pain experienced across all cycles of paclitaxel. Measured by the patient reported daily pain score from days 1 to 5 during all 4 cycles of paclitaxel chemotherapy. Bone pain is measured on a scale ranging from 0-10, 0 being no pain and 10 being the worst possible pain.
Patient health-related quality of life | Through study completion, average of 12 weeks
  Patient Health-Related Quality of Life (HR-QoL) based on the EuroQol 5 Dimension 5 Level (EQ-5D-5L) questionnaire.
Rates of completion of 4 cycles of paclitaxel | Through study completion, average of 12 weeks
  Rates of completion of 4 cycles of paclitaxel chemotherapy within 7 weeks (days 1 cycle 5 to day 1 cycle 8 of chemotherapy)
Dose-intensity of paclitaxel chemotherapy | Through study completion, average of 12 weeks
  Dose intensity of paclitaxel (mg/m2/wk) chemotherapy. Dose intensity is a measure of a dose delay/dose reduction and premature chemotherapy discontinuation.
Incidence of febrile neutropenia/neutropenia | Through study completion, average of 12 weeks
  Incidences of febrile neutropenia/neutropenia will be collected using pretreatment bloodwork that is routinely performed before each chemotherapy cycle. For this study, febrile neutropenia (FN) is defined as a one-time oral temperature greater or equal to 38.3 degrees Celsius (approximately 100.9 Fahrenheit) or a sustained temperature equal or greater than 38 degrees Celsius for 1 or more hours in a patient who has an absolute neutrophil count of less than 500 cells/microliter or an absolute neutrophil count expected to decrease to less than 500 cells/microliter within a 48-hour period.
Incidence of treatment-related hospitalizations/ER visits | Through study completion, average of 12 weeks
  The number of treatment-related hospitalizations and emergency room visits that occur from the start of paclitaxel chemotherapy to 1 month after the last paclitaxel chemotherapy cycle
Healthcare resource utilization: Emergency Room Visits | Through study completion, average of 12 weeks
  The number of emergency room visits that occur will be collected.
Healthcare resource utilization: Planned and Unplanned Provider Visits | Through study completion, average of 12 weeks
  The number of planned and unplanned provider clinic visits, including visits to stretcher bay will be collected.
Healthcare resource utilization: Phone Calls and Emails | Through study completion, average of 12 weeks
  The number of phone calls and emails to patient support line provider (reported by the patient) will be collected.
Cost-effectiveness ratios | Through study completion, average of 12 weeks
  There will be a cost-utility analysis comparing the differences in cost and quality-adjusted life years (QALY) between omitting G-CSF and standard G-CSF use. The statistical analysis will be conducted in accordance with current guidelines for clinical and cost-effectiveness analysis alongside randomized clinical trials (RCTs). Health utility values will be derived from EQ-5D-5L scores using the published mapping algorithm.
Incidence of chemotherapy-related mortality | Through study completion, average of 12 weeks
  Deaths from start of chemotherapy to one month after completion of last chemotherapy cycle
Rate of secondary G-CSF or antibiotic use | Through study completion, average of 12 weeks
  Rates of added G-CSF use for both randomization arms will be collected. As well as the addition of antibiotic use.

CONTACTS AND LOCATIONS:
Overall Officials: Xinni Song, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (3):
- Canada (3):
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Lakeridge Health, Oshawa, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario

REFERENCES:
- See also: The Rethinking Clinical Trials (REaCT) website — https://react.ohri.ca/